CLINICAL TRIAL: NCT00232726
Title: A Non-Randomised, Multicentre, Phase II Clinical Study of CP-4055 in Chemotherapy-Naïve Patients With Metastatic Malignant Melanoma
Brief Title: Clinical Study of Previously Untreated Patients With Malignant Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Clavis Pharma (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP4055-201
Record Dates: First submitted 2005-10-04; First posted 2005-10-05 (Estimated); Last update posted 2007-07-10 (Estimated); Status verified 2007-07

CONDITIONS: Malignant Melanoma; Neoplasm Metastasis
Keywords: Malignant melanoma; CP-4055; Chemotherapy-naïve patients; Phase II; Chemotherapy-naive patients; Metastatic malignant melanoma
MeSH Terms: conditions — Melanoma; Neoplasm Metastasis | interventions — 5'-oleoyl cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: CP-4055 (ELACYT)

SUMMARY:
Previously untreated patients with malignant melanoma receive a new chemotherapy drug currently under development. CP-4055 is given intravenously on days 1-5 every four weeks until complete response or disease progression.

DETAILED DESCRIPTION:
This is an international multicentre phase II clinical study conducted in the USA and Europe. Previously untreated patients over 18 years, with metastatic malignant melanoma are eligible for inclusion if they fulfil all inclusion- and exclusion criteria. 16 or 42 patients will be enrolled in Pittsburgh USA, Lund Sweden and Oslo Norway.

The new development drug CP-4055 is administered for five consecutive days (Day 1 to 5) in a 4 week schedule (one cycle). The dose is 200 mg/m2/day.

A patient will continue treatment until complete response or until (s)he is withdrawn from the Clinical Study because of disease progression, unacceptable toxicity or any other reason described in the clinical study protocol.

Efficacy is assessed at baseline and end of every second cycle with CT or MRI.

Safety assessments are done at each visit. Blood samples are taken and haematological and biochemical parameters are assessed for safety.

Any adverse events are recorded and reported.

The clinical study has been approved by the relevant Independent Ethical Committees/Institutional Review Boards and Concerned Regulatory Authority as appropriate. It is conducted according to ICH Good Clinical Practice, the Declaration of Helsinki, and applicable national law and regulations.

Patients who give an additional consent will have two additional, and not mandatory, procedures performed:

* Biopsy (tissue sample) from particular tumours (taken only at baseline for identification of tumour genes)
* Serum samples (from blood drawn at baseline and at end of the cycle 2 for protein sequences analyses, proteomics)

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically or cytologically confirmed stage IV or unresectable stage III non-ocular malignant melanoma who have not undergone prior chemotherapy for the treatment of melanoma (chemotherapy-naïve)
* Measurable disease according to Response Criteria in Solid Tumours (RECIST)
* Performance Status 0 - 2 according to ECOG (Eastern Cooperative Oncology Group) Performance Status
* Age 18 years or more
* Life expectancy > 3 months
* Signed informed consent
* Adequate haematological and biological functions:

  * Bone marrow function:

    1. Neutrophils ≥ 1.5 x 10^9/L
    2. Platelets ≥ 100 x 10^9/L
    3. Hemoglobin (Hb) ≥ 10 g/dL
  * Hepatic function:

    1. AST/ALT ≤ 2.5 times institutional upper limit of normal (ULN). If liver metastases, ≤ 5 times institutional ULN.
    2. Serum bilirubin and alkaline phosphatase ≤ 1.5 times institutional ULN
  * Renal function:

    * Creatinine ≤ 1.5 times institutional ULN

Exclusion Criteria:

* Known brain metastases
* Diagnosis of ocular malignant melanoma
* Radiotherapy to more than 30% of bone marrow
* Participation in another therapeutic clinical study within 30 days of enrolment or during this clinical study
* Prior immunotherapy and/or chemotherapy for the treatment of melanoma
* Requirement of concomitant treatment with a non-permitted medication:

  * Alternative drugs
  * High doses of vitamins
* History of allergic reactions to Ara-C or egg
* Presence of any serious concomitant systemic disorders incompatible with the clinical study (e.g. uncontrolled intercurrent illness including ongoing or active infection)
* Presence of any significant central nervous system or psychiatric disorder(s) that would hamper the patient's compliance
* Pregnancy, breastfeeding, or absence of adequate contraception for both male and female fertile patients
* Known positive status for HIV and/or hepatitis B or C
* Drug and/or alcohol abuse
* Any reason why, in the Investigator's opinion, the patient should not participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2005-09; Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Objective tumour response

SECONDARY OUTCOMES:
Time to progression
Duration of tumour response
Safety and tolerability of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Svein Dueland, MD, Ph.D, Principal Investigator — The Norwegian Radium Hospital, Montebello, NO-0310 Oslo, Norway
Locations (3):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States
- The Norwegian Radium Hospital, Oslo, Norway
- University Hospital, Lund, Sweden

REFERENCES:
- See also: Sponsor's home page — http://www.clavispharma.com